CLINICAL TRIAL: NCT07049471
Title: The Effect of Swallowing Exercise and Maneuver Program For Older Adults With Dysphagia in Nursing Home
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Direktorat Riset dan Pengabdian Masyarakat Universitas Indonesia (Unknown)
Responsible Party: Principal Investigator, Etty Rekawati, Principal Investigator of the Clinical Trial, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NKB-215/UN2.RST/HKP.05.00/2024; NKB-215/UN2.RST/HKP.05.00/2024 (Other Grant/Funding Number: Directorate of Research and Development, Universitas Indonesia under Hibah PUTI 2024)
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Oropharyngeal Dysphagia; Swallowing Disorders; Frailty-related Dysphagia; Nursing Homes
Keywords: Oropharyngeal Dysphagia; older adult; nursing home; swallowing
MeSH Terms: conditions — Deglutition Disorders | interventions — Aging

STUDY DESIGN:
Intervention Model Description: This study used a randomized, parallel-group design involving two arms: an intervention group receiving a structured swallowing exercise and maneuver program, and a control group receiving standard care. Participants were randomly assigned using a simple random sampling technique. The intervention was administered three times daily for six weeks. Outcomes were compared between groups to evaluate the effectiveness of the intervention on swallowing function in older adults with oropharyngeal dysphagia living in a nursing home.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swallowing Exercise and Maneuver Group (Experimental): Participants in this arm received a structured swallowing exercise and maneuver program consisting of four techniques: Masako Maneuver, Chin Tuck Against Resistance (CTAR), Supraglottic Swallow, and Super-Supraglottic Swallow. The exercises were administered by nurses using a video-guided protocol, three times daily before meals for six weeks. The program was designed to improve pharyngeal muscle strength and enhance airway protection during swallowing.
  Interventions: Behavioral: Swallowing Exercise and Maneuver Program for Older Adults with Dysphagia
- Standard Care Group (No Intervention): Participants in this arm received standard care for dysphagia, which involved upright sitting positioning during meals without any structured swallowing exercises or maneuvers. No additional behavioral interventions were provided during the study period.

INTERVENTIONS:
Behavioral: Swallowing Exercise and Maneuver Program for Older Adults with Dysphagia — The intervention is a structured swallowing exercise and maneuver program designed specifically for older adults with oropharyngeal dysphagia in nursing homes. It combines four evidence-based techniques: Masako Maneuver, Chin Tuck Against Resistance (CTAR), Supraglottic Swallow, and Super-Supraglottic Swallow. The program was delivered by nurses using video-guided instructions and was conducted three times daily before meals for six weeks. Unlike interventions targeting post-stroke dysphagia, this program focuses on non-stroke-related swallowing difficulties in frail elderly populations residing in long-term care facilities.
  Arms: Swallowing Exercise and Maneuver Group

SUMMARY:
This clinical trial aimed to evaluate the effectiveness of a structured swallowing exercise and maneuver program for older adults with dysphagia living in a nursing home. Dysphagia, or difficulty in swallowing, is common in elderly populations and may lead to malnutrition, dehydration, and aspiration pneumonia.

In this study, 72 participants aged 60 years and older were randomly assigned to either an intervention group or a control group. The intervention group received a combined swallowing exercise and maneuver program-including Masako Maneuver, Chin Tuck Against Resistance, Supraglottic Swallow, and Super-Supraglottic Swallow-performed three times daily before meals over a six-week period. The control group received standard care, including upright sitting posture during meals.

Swallowing ability was measured using the EAT-10 questionnaire. The intervention group showed significant improvement in swallowing scores, while no meaningful changes were observed in the control group. This study suggests that nurse-led swallowing exercises can be a safe, simple, and effective strategy to improve swallowing function and quality of life in older adults living in long-term care settings.

DETAILED DESCRIPTION:
Oropharyngeal dysphagia is a prevalent condition among older adults, particularly in institutionalized settings such as nursing homes. It is often underdiagnosed, misattributed to normal aging, and leads to serious complications including aspiration pneumonia, malnutrition, dehydration, and diminished quality of life. Despite its high burden, non-pharmacological interventions tailored to this population in Indonesia remain limited.

This randomized controlled trial was designed to assess the effectiveness of a structured swallowing exercise and maneuver program for older adults with dysphagia in a long-term care facility. The intervention integrated both pharyngeal element-based exercises (Masako Maneuver and Chin Tuck Against Resistance) and behavioral-based exercises (Supraglottic Swallow and Super-Supraglottic Swallow). These exercises were delivered as a video-guided program and administered three times per day before meals over six weeks by trained nursing staff.

Participants were randomly assigned to intervention and control groups using a simple random sampling method. The control group received standard care without swallowing exercises. Outcomes were measured using the Eating Assessment Tool-10 (EAT-10), a validated instrument for identifying clinically significant swallowing problems.

This study aimed to provide empirical evidence for the use of structured, nurse-delivered swallowing training as an effective and feasible approach to managing dysphagia among the elderly in nursing homes. It also explored the potential for routine implementation and integration into geriatric nursing practice across similar institutional care settings.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years or older
* experiencing swallowing difficulties as assessed by the Eating Assessment Tool-10 (EAT-10)
* having no history of neurological disease
* possessing adequate communication abilities
* and being capable of performing daily activities either independently or with partial assistance

Exclusion Criteria:

* individuals with dermatological conditions in the anterior neck region, hypertension, orofacial pain such as trigeminal neuropathy or toothache, as well as those with significant malocclusion or facial asymmetry

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Swallowing Function Measured by EAT-10 Score | Baseline (Day 0) and Week 6 (Post-intervention)
  Swallowing function is assessed using the Eating Assessment Tool-10 (EAT-10), a validated 10-item self-report questionnaire for identifying symptoms of dysphagia. Each item is scored from 0 (no problem) to 4 (severe problem), with a total possible score ranging from 0 to 40. A score of 3 or more indicates clinically significant dysphagia. The primary outcome is the change in EAT-10 scores from baseline (prior to intervention) to the end of the 6-week intervention period. A decrease in score reflects improvement in swallowing function.
Change in Swallowing Function as Measured by EAT-10 Score | Baseline and 6 weeks after intervention initiation
  Swallowing function was assessed using the Eating Assessment Tool-10 (EAT-10), a validated 10-item questionnaire designed to identify symptoms of dysphagia. Each item is scored on a 5-point Likert scale (0-4), with total scores ranging from 0 to 40. A score ≥3 indicates clinically significant swallowing difficulty. The primary outcome is the change in total EAT-10 score from baseline (pre-intervention) to the end of the 6-week intervention period. A greater reduction in the EAT-10 score indicates an improvement in swallowing function.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing Universitas Indonesia, Depok, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be shared upon reasonable request for academic or scientific purposes.
Supporting Information: Study Protocol